CLINICAL TRIAL: NCT01155830
Title: Inflammatory Cytokine Quantification in Infants With Documented Sepsis, Congenital Diaphragmatic Hernia and/or ECMO Therapy
Brief Title: Inflammatory Cytokine Quantification in Infants
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Dr. Donald Null, University of Utah
Other Study IDs: 39121
Record Dates: First submitted 2010-06-22; First posted 2010-07-02 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2014-12

CONDITIONS: Sepsis; Congenital Diaphragmatic Hernia; Neonatal Cardiopulmonary Failure
Keywords: inflammatory cytokines; extracorporeal membrane oxygenation; ECMO
MeSH Terms: conditions — Sepsis; Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Infants with CHD: Infants with Congenital Diaphragmatic Hernia (CHD)
- Infants with sepsis: Infants who are culture positive for sepsis and require vasopressor support
- Infants treated with ECMO: Infants suffering cardiopulmonary failure significant enough to require heart/lung bypass treatment with extracorporeal membrane oxygenation (ECMO)

SUMMARY:
This study proposes to quantify inflammatory cytokine profiles in three neonatal disease states, namely, neonatal sepsis, infants with a congenital diaphragmatic hernia defect, and infants suffering cardiopulmonary failure significant enough to require heart/lung bypass treatment with extracorporeal membrane oxygenation (ECMO).

DETAILED DESCRIPTION:
Very small blood samples (500 microliters) will be collected serially in these patients and analyzed with current cytokine array technology. A convenience sample of 60 patients, 20 with each of these diagnoses, will be collected over a 2 year period. These data will provide baseline information for possible therapeutic intervention with agents that enhance or suppress specific mediators, or adjust mediator balance to promote patient healing.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 34 weeks,
* Indwelling vascular catheter available for blood draws,
* Documented culture positive sepsis on vasopressors , and/or
* Congenital diaphragmatic hernia (CDH), and/or
* ECMO therapy

Exclusion Criteria:

* Other major congenital anomalies
* Lack of parental consent

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admitted into the NICU at the University of Utah Health Sciences Centers and Primary Children's Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Null, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infants With CHD | Infants With Sepsis | Infants Treated With ECMO
Started | 0 | 0 | 21
Completed | 0 | 0 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infants With CHD | Infants With Sepsis | Infants Treated With ECMO | Total
Number analyzed (Participants) | 0 | 0 | 21 | 21
Age, Categorical [Number; unit: participants]
  <=18 years |  |  | 21 | 21
  Between 18 and 65 years |  |  | 0 | 0
  >=65 years |  |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] |  |  | 1 (1) | 1 (1)
Gender [Number; unit: participants]
  Female |  |  | 8 | 8
  Male |  |  | 13 | 13
Region of Enrollment [Number; unit: participants]
  United States |  |  | 21 | 21

OUTCOME MEASURES:

1. Primary Outcome: TNF-alpha, Baseline
Description: This study will quantify inflammatory cytokine profiles in three neonatal disease states, namely, neonatal sepsis with cardiovascular instability, infants with a congenital diaphragmatic hernia defect, and infants suffering cardiopulmonary failure significant enough to require heart/lung bypass treatment with extracorporeal membrane oxygenation (ECMO).
Time Frame: Baseline
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Infants With CHD | Infants With Sepsis | Infants Treated With ECMO
Number analyzed (Participants) | 0 | 0 | 21
pg/mL |  |  | 8.88 (4.58)

2. Secondary Outcome: TNF-alpha, Maximum
Description: as for outcome 1
Time Frame: up to 2 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Infants With CHD | Infants With Sepsis | Infants Treated With ECMO
Number analyzed (Participants) | 0 | 0 | 21
pg/mL |  |  | 33.1 (9.373)

ADVERSE EVENTS:
Arm/Group | Infants With CHD | Infants With Sepsis | Infants Treated With ECMO
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/21
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes